CLINICAL TRIAL: NCT05438212
Title: A Randomized Phase III Trial of Pre-Operative Compared to Post-Operative Stereotactic Radiosurgery in Patients With Resectable Brain Metastases
Brief Title: Comparing the Addition of Radiation Either Before or After Surgery for Patients With Brain Metastases
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BN012; NCI-2022-04804 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN012 (Other: NRG Oncology); NRG-BN012 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (surgery, stereotactic radiosurgery) (Active Comparator): Patients undergo surgery per standard of care. Within 10-30 days after surgery, patients undergo stereotactic radiosurgery for 1 fraction.
  Interventions: Procedure: Brain Surgery; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery
- Arm II (stereotactic radiosurgery, surgery) (Experimental): Within 7 days before surgery, patients undergo stereotactic radiosurgery for 1 fraction. Patients undergo surgery per standard of care.
  Interventions: Procedure: Brain Surgery; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Procedure: Brain Surgery — Undergo surgery per standard of care
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Radiosurgery — Undergo stereotactic radiosurgery
  Other Names: SRS; Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery

SUMMARY:
This phase III trial compares the usual treatment of surgery after stereotactic radiosurgery (SRS) to receiving SRS before surgery in treating patients with cancer that has spread to the brain (brain metastases). Stereotactic radiosurgery is a type of radiation therapy that delivers a high dose of radiation to target tumors and minimizes effect on normal surrounding brain tissue. The combination of surgery and radiation may stop the tumor from growing for a few months or longer and may reduce symptoms of brain metastases. This study investigates whether treating with SRS before surgery may be better than SRS after surgery in reducing the possibility of the tumor coming back, reducing or preventing the cancer from spreading to other areas of the brain and reducing the risk of scarring on the brain from radiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the time to composite adverse endpoint (CAE) (defined as: 1) local tumor progression within the surgical bed; and/or 2) adverse radiation effect [ARE], the imaging correlate of post-stereotactic radiosurgery [SRS] radiation necrosis; and/or 3) nodular meningeal disease [nMD]) is improved in patients treated with pre-resection SRS to the intact lesion versus those treated with post-resection SRS.

SECONDARY OBJECTIVES:

I. To assess the trajectory of symptom burden in patients treated with pre-resection SRS to the intact lesion versus those treated to the post-resection surgical cavity as measured by MD Anderson Symptom Inventory for brain tumor (MDASI-BT).

II. To determine whether there is improved overall survival (OS) in patients with resected brain metastases who undergo pre-resection SRS compared to patients who receive post-resection SRS.

III. To compare rates of ARE, the imaging correlate of radiation necrosis, in patients who receive pre-resection SRS to patients who receive post-resection SRS.

IV. To determine whether there is increased time to whole brain radiotherapy (WBRT) in patients who receive pre-resection SRS compared to patients who receive post-resection SRS.

V. To assess the trajectory of neuro-cognitive function in patients treated with pre-resection SRS to the intact lesion versus those treated to the post-resection surgical cavity as measured by the Montreal Cognitive Assessment (MoCA).

VI. To compare rates of nodular meningeal disease in patients who receive pre-resection SRS to patients who receive post-resection SRS.

VII. To compare rates of local recurrence in the resection cavity for patients who receive pre-resection SRS to patients who receive post-resection SRS.

VIII. To compare rates of local recurrence of intact, non-index metastases treated with SRS.

IX. To compare rates of distant brain failure in patients who receive pre-resection SRS to patients who receive post-resection SRS.

X. To assess toxicity in the two treatment arms.

EXPLORATORY OBJECTIVE:

I. To explore if the type of surgical resection (piece-meal versus [vs.] en-bloc) may be associated with the rate of nodular meningeal disease.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo surgery per standard of care. Within 10-30 days after surgery, patients undergo stereotactic radiosurgery for 1 fraction.

ARM II: Within 7 days before surgery, patients undergo stereotactic radiosurgery for 1 fraction. Patients undergo surgery per standard of care.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for additional 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic confirmation of 1-4 brain metastases, one of which requires resection, as defined by magnetic resonance imaging (MRI) with contrast obtained within 14 days prior to registration

  * The maximum diameter of the lesion to be resected on the post-contrast MRI, as measured on any orthogonal plane (axial, sagittal, coronal), must measure >= 2.0 cm and =< 5.0 cm.
  * The maximum diameter of any lesions which will not be resected must be =< 4.0 cm in maximum diameter
* Known active or history of invasive non-central nervous system (CNS) primary cancer based on documented pathologic diagnosis within the past 3 years
* All brain metastases must be located >= 5 mm from the optic chiasm and outside the brainstem
* Patient is able to medically tolerate surgery and SRS
* Lesions chosen for surgical therapy must be deemed appropriate targets for safe, gross total resection by the treating surgeon
* History/physical examination within 14 days prior to registration
* Age >= 18
* Karnofsky performance status (KPS) >= 60 within 14 days prior to registration
* A negative urine or serum pregnancy test (in persons of childbearing potential) within =< 14 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal
* Participants who are sexually active must agree to use medically acceptable forms of contraception during treatment on this study to prevent pregnancy
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Prior cranial radiotherapy, including whole brain radiotherapy, or SRS to the resection site

  * Note: The index lesion to be resected cannot have been previously treated with SRS (i.e. repeat radiosurgery to the same location/lesion is not allowed on this protocol). Previous SRS to other lesions is allowed
* Evidence of leptomeningeal disease (LMD)

  * Note: For the purposes of exclusion, LMD is a clinical diagnosis, defined as positive cerebrospinal fluid (CSF) cytology and/or unequivocal radiologic or clinical evidence of leptomeningeal involvement. Patients with leptomeningeal symptoms in the setting of leptomeningeal enhancement by imaging (MRI) would be considered to have LMD even in the absence of positive CSF cytology. In contrast, an asymptomatic or minimally symptomatic patient with mild or nonspecific leptomeningeal enhancement (MRI) would not be considered to have LMD. In that patient, CSF sampling is not required to formally exclude LMD, but can be performed at the investigator's discretion based on level of clinical suspicion
* Any medical conditions which would make this protocol unreasonably hazardous, including, but not limited to: contraindications to general endotracheal anesthesia; intracranial surgery; and stereotactic radiosurgery
* Primary histology of germ cell tumor, small cell carcinoma or lymphoma
* More than one brain metastasis planned for resection
* Inability to undergo MRI with contrast
* Planned administration of cytotoxic chemotherapy or tyrosine/multi-kinase inhibitors within the 3 days prior to, the day of, or within 3 days after the completion of SRS

  * Note: chemotherapy and immunotherapy outside of this window are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2027-03-16 (Estimated); Study Completion 2027-03-16 (Estimated)

PRIMARY OUTCOMES:
Time to composite adverse endpoint (CAE) | Time from surgery (with the post-operative MRI as the 'baseline' for purposes of disease assessment) to local tumor progression (within the surgical bed), nodular meningeal disease, or radiation necrosis, whichever occurs first, assessed up to 4 years
  Analysis for this endpoint will consist of testing the cause-specific hazard ratio in a Cox proportional hazards model.

SECONDARY OUTCOMES:
Overall survival (OS) | Time from randomization to death due to any cause, assessed up to 4 years
  Analysis for this endpoint will consist of estimation of the OS distribution of each treatment arm via the Kaplan-Meier method and a stratified log-rank test.
Rate of local tumor progression | Up to 4 years
  The time origin for these imaging-based endpoints will be time of surgery (with the post-operative magnetic resonance imaging [MRI] as the 'baseline' for purposes of disease assessment). These analyses will involve estimating the cumulative incidence function of local progression, radiation necrosis, nodular meningeal disease, and distant brain failures in the presence of competing event of deaths. The Gray's test will be used to evaluate the difference in the distribution of local progression between treatment arms.
Rate of radiation necrosis | Up to 4 years
  The time origin for these imaging-based endpoints will be time of surgery (with the post-operative MRI as the 'baseline' for purposes of disease assessment). These analyses will involve estimating the cumulative incidence function of local progression, radiation necrosis, nodular meningeal disease, and distant brain failures in the presence of competing event of deaths. The Gray's test will be used to evaluate the difference in the distribution of radiation necrosis between treatment arms.
Rate of nodular meningeal disease | Up to 4 years
  The time origin for these imaging-based endpoints will be time of surgery (with the post-operative MRI as the 'baseline' for purposes of disease assessment). These analyses will involve estimating the cumulative incidence function of local progression, radiation necrosis, nodular meningeal disease, and distant brain failures in the presence of competing event of deaths. The Gray's test will be used to evaluate the difference in the distribution of nodular meningeal disease between treatment arms.
Rate of distant brain failures | Up to 4 years
  The time origin for these imaging-based endpoints will be time of surgery (with the post-operative MRI as the 'baseline' for purposes of disease assessment). These analyses will involve estimating the cumulative incidence function of local progression, radiation necrosis, nodular meningeal disease, and distant brain failures in the presence of competing event of deaths. The Gray's test will be used to evaluate the difference in the distribution of distant brain failures between treatment arms.
Frequency of adverse events (AEs) | Up to 4 years
  AEs will be graded according to Common Terminology Criteria for Adverse Events version 5.0. Comprehensive summaries of all AEs by treatment arm will be generated and examined. Counts and frequencies of worst (highest score) AE per patient will be presented overall and by AE type category, separately by assigned treatment group. The proportion of patients with at least one grade 3 or higher AE will be compared between treatment arms. Any frequencies to be tested will be evaluated using the chi-square or exact test as appropriate, with two-sided significance level 0.05.
Change in MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT) | Baseline up to 2 years after surgery
  Will implement mixed effects models for repeated measures to evaluate the MDASI-BT scores longitudinally.
Change in cognitive function | Baseline up to 2 years after surgery
  Measured by Montreal Cognitive Assessment (MoCA). Will implement mixed effects models for repeated measures to evaluate the MoCA scores longitudinally.

OTHER OUTCOMES:
Type of surgical resection | Up to 4 years
  Will compare if the type of surgical resection (piece-meal vs. en-bloc) may be associated with the rate of nodular meningeal disease. The competing risk approach by Gray (Gray 1988) will be used to compare the cumulative incidences of nMD by surgical type, where death prior to nMD will be treated as a competing risk event. This analysis will only include patients who undergo surgical resections at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart H Burri, Principal Investigator — NRG Oncology
Locations (215):
- United States (207):
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Advocate Outpatient Center - Aurora, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - UM Capital Region Medical Center, Largo, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The New York Hospital Medical Center of Queens, Flushing, New York
  - Northern Westchester Hospital, Mount Kisco, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Good Samaritan University Hospital, West Islip, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Henrico Doctor's Hospital, Richmond, Virginia
  - CJW Medical Center - Johnston-Willis Campus, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (3):
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
- Japan (5):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Gunma University Hospital, Gunma, Maebashi
  - Kyoto University Hospital, Kyoto
  - Nagoya University Hospital, Showa-Ku Nagoya
  - National Cancer Center Hospital, Tokyo

REFERENCES:
- [Derived] Prabhu RS, Akinyelu T, Vaslow ZK, Matsui JK, Haghighi N, Dan T, Mishra MV, Murphy ES, Boyles S, Perlow HK, Palmer JD, Udovicich C, Patel TR, Wardak Z, Woodworth GF, Ksendzovsky A, Yang K, Chao ST, Asher AL, Burri SH. Single-Fraction Versus Fractionated Preoperative Radiosurgery for Resected Brain Metastases: A PROPS-BM International Multicenter Cohort Study. Int J Radiat Oncol Biol Phys. 2024 Mar 1;118(3):650-661. doi: 10.1016/j.ijrobp.2023.09.012. Epub 2023 Sep 16. PMID 37717787
- [Derived] Prabhu RS, Akinyelu T, Vaslow ZK, Matsui JK, Haghighi N, Dan T, Mishra MV, Murphy ES, Boyles S, Perlow HK, Palmer JD, Udovicich C, Patel TR, Wardak Z, Woodworth GF, Ksendzovsky A, Yang K, Chao ST, Asher AL, Burri SH. Risk Factors for Progression and Toxic Effects After Preoperative Stereotactic Radiosurgery for Patients With Resected Brain Metastases. JAMA Oncol. 2023 Aug 1;9(8):1066-1073. doi: 10.1001/jamaoncol.2023.1629. PMID 37289451